CLINICAL TRIAL: NCT02770716
Title: A Multi-Center, Randomized, Placebo Controlled, Double-Blind Study to Confirm Efficacy and Safety of Terlipressin in Subjects With Hepatorenal Syndrome Type 1 (The CONFIRM Study)
Brief Title: Study To Confirm Efficacy and Safety of Terlipressin in Hepatorenal Syndrome (HRS) Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK19013058
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Results first posted 2022-08-18 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hepatorenal Syndrome
Keywords: Type 1
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Terlipressin (Experimental): Participants receive terlipressin intravenously as a bolus injection, followed by a saline flush. Dose, duration, retreatment and/or discontinuation may be modified by the investigator, per protocol.
  Interventions: Drug: Terlipressin
- Placebo (Placebo Comparator): Participants receive matching placebo intravenously as a bolus injection, followed by a saline flush. Dose, duration, retreatment and/or discontinuation may be modified by the investigator, per protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Terlipressin — Terlipressin solution for injection
  Arms: Terlipressin
Other: Placebo — Matching placebo solution for injection
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
This study is to treat adult patients with hepatorenal syndrome (HRS) Type 1.

Out of every three participants, two will receive terlipressin and one will receive placebo.

Assignments will be made randomly.

DETAILED DESCRIPTION:
The primary objective of this trial is to confirm the efficacy and safety of intravenous terlipressin versus placebo in the treatment of adult subjects with hepatorenal syndrome (HRS) Type 1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by participant or legally authorized representative
* Cirrhosis and ascites
* Rapidly progressive worsening in renal function to a serum creatinine (SCr) at least 2.25 mg/dL and meeting a trajectory for SCr to double over 2 weeks
* No sustained improvement in renal function (less than 20% decrease in SCr and SCr at least 2.25 mg/dL) at least 48 hours after diuretic withdrawal and the beginning of plasma volume expansion with albumin
* Discontinues midodrine and octreotide before randomization if applicable

Exclusion Criteria:

* Serum creatinine level greater than 7.0 mg/dL
* At least 1 event of large volume paracentesis (LVP) at least 4 L within 2 days of randomization
* Sepsis and/or uncontrolled bacterial infection
* Less than 2 days anti-infective therapy for documented or suspected infection
* Shock
* Being treatment with or exposure to nephrotoxic agents, nonsteroidal anti-inflammatory drugs, or significant radiographic contrast agents (within the last 4 weeks)
* Estimated life expectancy of less than 3 days
* Superimposed acute liver injury due to drugs, dietary supplements, herbal preparations, viral hepatitis, or toxins, with the exception of acute alcoholic hepatitis
* Proteinuria greater than 500 mg/day
* Evidence of obstructive uropathy or parenchymal renal disease on ultrasound or other imaging
* Tubular epithelial casts, heme granular casts, hematuria or microhematuria (greater than 50 red blood cells per high power field in the absence of recent catheterization) on urinalysis
* Pregnancy; all women of child-bearing age and potential must have a negative pregnancy test
* Cardiovascular disease judged by the investigator to be severe
* Current or recent renal replacement therapy (RRT) within the past 4 weeks
* Participation in other clinical research involving investigational medicinal products within 30 days of randomization
* Transjugular intrahepatic portosystemic shunt (TIPS) within 30 days of randomization
* Use of vasopressors for at least 3 consecutive days within the 14-day screening period - patients receiving any vasopressor other than midodrine and octreotide within 24 hours of qualifying SCr are also excluded, ie, a 24-hour washout is required prior to enrollment
* Known allergy or sensitivity to terlipressin or another component of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Lead, Study Director — Mallinckrodt
Locations (64):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Mayo Clinic - AZ, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - USC Healthcare, Los Angeles, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - UCLA Medical Center, San Diego, California
  - Southern California Research Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic - FL, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Hospital Transplant, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - MN, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - NYU Langone Health, New York, New York
  - Weil Cornell Medical College, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Case Western Reserve Transplant, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Drexel University, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson University, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Parkland Health and Hospital System, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor Scott and White All Saints Medical Center, Fort Worth, Texas
  - Baylor College of Medicine (St. Luke's), Houston, Texas
  - Methodist Center for Liver Disease and Transplantation, Houston, Texas
  - Methodist Transplant Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center/Univ. of Washington, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Canada (5):
  - Vancouver General Hospital, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Ottawa Hospital, Ottawa, Ontario
  - University of Toronto 9N/983 Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal
  - Centre Hospitalier de l'Université de Montréal, Québec

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT02770716) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Rockey DC, Gordon F, Thuluvath PJ, Victor D, Kemmer N, Cardoza S, Jamil K, Frederick RT. Terlipressin for Hepatorenal Syndrome in Patients With Early-Stage Acute-on-Chronic Liver Failure. Liver Int. 2025 Dec;45(12):e70399. doi: 10.1111/liv.70399. PMID 41200852
- [Derived] Bajaj JS, Kwo P, Pappas SC, O'Leary JG, Jamil K, Cardoza S, Wong F. Bradycardia and Other Arrhythmias in Patients With Hepatorenal Syndrome-Acute Kidney Injury Following Terlipressin Treatment: A Pooled Analysis of Three North American Phase III Clinical Studies. Aliment Pharmacol Ther. 2025 Dec;62(11-12):1192-1201. doi: 10.1111/apt.70297. Epub 2025 Jul 24. PMID 40704461
- [Derived] Mujtaba MA, Gamilla-Crudo AK, Merwat SN, Hussain SA, Kueht M, Karim A, Khattak MW, Rooney PJ, Jamil K. Terlipressin in combination with albumin as a therapy for hepatorenal syndrome in patients aged 65 years or older. Ann Hepatol. 2023 Sep-Oct;28(5):101126. doi: 10.1016/j.aohep.2023.101126. Epub 2023 Jun 10. PMID 37302573
- [Derived] Velez JCQ, Wong F, Reddy KR, Sanyal AJ, Vargas HE, Curry MP, Gonzalez SA, Pappas SC, Jamil K. The Effect of Terlipressin on Renal Replacement Therapy in Patients with Hepatorenal Syndrome. Kidney360. 2023 Aug 1;4(8):1030-1038. doi: 10.34067/KID.0000000000000132. Epub 2023 May 5. PMID 37143199
- [Derived] Curry MP, Vargas HE, Befeler AS, Pyrsopoulos NT, Patwardhan VR, Jamil K. Early treatment with terlipressin in patients with hepatorenal syndrome yields improved clinical outcomes in North American studies. Hepatol Commun. 2023 Jan 3;7(1):e1307. doi: 10.1097/01.HC9.0000897228.91307.0c. eCollection 2023 Jan 1. PMID 36633470
- [Derived] Wong F, Pappas SC, Curry MP, Reddy KR, Rubin RA, Porayko MK, Gonzalez SA, Mumtaz K, Lim N, Simonetto DA, Sharma P, Sanyal AJ, Mayo MJ, Frederick RT, Escalante S, Jamil K; CONFIRM Study Investigators. Terlipressin plus Albumin for the Treatment of Type 1 Hepatorenal Syndrome. N Engl J Med. 2021 Mar 4;384(9):818-828. doi: 10.1056/NEJMoa2008290. PMID 33657294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 60 active sites in the United States and Canada
Period: Overall Study
Arm/Group | Terlipressin | Placebo
Started | 199 | 101
Intent to Treat (ITT) | 199 | 101
Safety Analysis Set (SAS) | 200 (One placebo participant received terlipressin as well, so is included in the terlipressin SAS) | 99 (One placebo participant did not receive any treatment, so was excluded from the SAS)
Systemic Inflammatory Response Syndrome (SIRS) Subgroup (SIRS subgroup included all participants from the ITT population who met the SIRS criteria.) | 84 | 48
Completed | 87 (ITT Completed Study through Follow-up / Day 90 Visit) | 52 (ITT Completed Study through Follow-up / Day 90 Visit)
Not Completed | 112 | 49
Not completed — Death | 101 | 45
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Various reasons | 6 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Terlipressin | Placebo | Total
Number analyzed (Participants) | 199 | 101 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.34) | 53.6 (11.83) | 53.8 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 42 | 121
  Male | 120 | 59 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 13 | 45
  Not Hispanic or Latino | 165 | 88 | 253
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 5 | 17
  White | 177 | 94 | 271
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 12 | 33
  United States | 178 | 89 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Verified HRS Reversal
Description: Defined as the percentage of participants with 2 consecutive SCr values ≤ 1.5 mg/dL at least 2 hours apart, while on treatment by Day 14 or discharge (on treatment defined as up to 24 hours after the final dose of study drug), per protocol.
Time Frame: within 15 Days
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 199 | 101
percentage of participants | 29.1 | 15.8

2. Primary Outcome: Percentage of Participants Who Were Viable (Per Protocol) for Inclusion in the Primary End Point Analysis
Description: Defined as the percentage of participants with verified HRS reversal who lived at least 10 days without RRT, and were otherwise viable (per protocol) for inclusion in the primary endpoint analysis
Time Frame: within 25 days
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 199 | 101
percentage of participants | 91.3 | 94.4

3. Secondary Outcome: Percentage of Participants With HRS Reversal
Description: Defined as the percentage of participants with a SCr value no more than 1.5 mg/dL by Day 14 or discharge, and were viable (per protocol) for inclusion in the secondary endpoint analysis
Time Frame: within 14 days
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 199 | 101
percentage of participants | 36.2 | 16.8

4. Secondary Outcome: Percentage of Participants With Durable HRS Reversal
Description: Defined as the percentage of participants maintaining HRS reversal without RRT to Day 30
Time Frame: Day 30
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 199 | 101
percentage of participants | 31.7 | 15.8

5. Secondary Outcome: Percentage pf Participants in the SIRS Subgroup With HRS Reversal
Description: Defined as the percentage of participants in the SIRS subgroup with HRS reversal by Day 14 or discharge
Time Frame: within 14 days
Population: ITT participants in the SIRS subgroup
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 84 | 48
percentage of participants | 33.3 | 6.3

6. Secondary Outcome: Percentage of Participants With Verified HRS Reversal Without HRS Recurrence by Day 30
Description: Defined as the percentage of participants who had achieved verified HRS reversal by Day 15 or discharge and did not revert to baseline measures by day 30
Time Frame: Day 30
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 199 | 101
percentage of participants | 24.1 | 15.8

ADVERSE EVENTS:
Time Frame: SAEs are collected in the safety analysis set (SAS) from informed consent to 30 days post-treatment; deaths are collected through study completion at 90 days from treatment start
Description: Participants experiencing multiple episodes of a given adverse event are counted once within each preferred term and within each system organ class.
Arm/Group | Terlipressin | Placebo
All-Cause Mortality (participants affected / at risk) | 101/200 | 45/99
Serious Adverse Events (participants affected / at risk) | 142/200 | 62/99
Other Adverse Events (participants affected / at risk) | 157/200 | 82/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terlipressin (N=200) | Placebo (N=99)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 11 (11) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 14 (14) | 8 (8)
Cirrhosis alcoholic (Hepatobiliary disorders) | 5 (5) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 8 (8) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 11 (11) | 10 (10)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 3 (3) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver transplant rejection (Immune system disorders) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 10 (11) | 0 (0)
Septic shock (Infections and infestations) | 7 (8) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Body temperature fluctuation (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Coma hepatic (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 9 (9) | 3 (4)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 4 (4) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)
Shock (Vascular disorders) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terlipressin (N=200) | Placebo (N=99)
Anaemia (Blood and lymphatic system disorders) | 13 (14) | 6 (6)
Bradycardia (Cardiac disorders) | 10 (11) | 0 (0)
Tachycardia (Cardiac disorders) | 10 (10) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 38 (46) | 5 (5)
Ascites (Gastrointestinal disorders) | 10 (10) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 26 (30) | 7 (7)
Nausea (Gastrointestinal disorders) | 32 (32) | 10 (10)
Vomiting (Gastrointestinal disorders) | 17 (17) | 9 (10)
Chest pain (General disorders) | 11 (11) | 3 (3)
Pyrexia (General disorders) | 4 (4) | 7 (8)
Urinary tract infection (Infections and infestations) | 6 (6) | 6 (6)
Fluid overload (Metabolism and nutrition disorders) | 15 (15) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (17) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 17 (19) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 4 (4)
Hypotension (Vascular disorders) | 16 (16) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02770716/Prot_SAP_001.pdf